CLINICAL TRIAL: NCT02683837
Title: A Prospective Randomized Study Evaluating Pupillometry Guided Remifentanil Administration in Pediatric Anesthesia
Brief Title: Pupillometry Guided Remifentanil Administration In Pediatric Anesthesia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal investigator left the institution
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Walid HABRE, Professor, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pupilloped
Record Dates: First submitted 2016-01-19; First posted 2016-02-17 (Estimated); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Anesthesia; Pain; Child
Keywords: Intraoperative Neurophysiological Monitoring; Reflex, Pupillary; remifentanil
MeSH Terms: conditions — Pain | interventions — Remifentanil; Sevoflurane

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard practice (Active Comparator): Remifentanil infusion guided by usual clinical signs (heart rate, blood pressure).
  Pupillometry blindly recorded. Anesthesia maintenance with sevoflurane.
  Interventions: Drug: Remifentanil; Drug: Sevoflurane
- Pupillometry (Experimental): Remifentanil infusion guided by changes in pupillary diameter. Anesthesia maintenance with sevoflurane.
  Interventions: Drug: Remifentanil; Device: Pupillometry; Drug: Sevoflurane

INTERVENTIONS:
Drug: Remifentanil
Device: Pupillometry — Pupillary diameter measured every 5 minutes
  Arms: Pupillometry
Drug: Sevoflurane — Administered to maintain a Bispectral Index between 40 and 60

SUMMARY:
The aim of this prospective randomized study is to evaluate the impact of peroperative pupillometry monitoring on per and post-operative opioid consumption in pediatric anesthesia. All patients are anesthetized with sevoflurane and remifentanil. In the intervention group, peroperative remifentanil infusion rate is guided by pupillometry. In the other group, remifentanil infusion rate is guided according to hemodynamic data.

ELIGIBILITY:
Inclusion Criteria:

* Children scheduled for a surgery lasting more than 90 minutes.

Exclusion Criteria:

* Contraindication to sevoflurane, to remifentanil or to morphine.
* Peripheral or central nerve block during and after surgery.
* Ophthalmological disease.
* Peroperative position with no acess to the head.
* Chronic use of medication interfering with pupillary diameter.
* Ambulatory surgery

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
peroperative remifentanil consumption | duration of surgery

SECONDARY OUTCOMES:
Morphine consumption | during the 24 hour post operative period
Incidence of morphine side effects | during the 24 hour post operative period
  Sedation, nausea, vomiting, pruritus, urinary retention
Pain scoring (verbal numerical scale) | during the 24 hour post operative period
Pain scoring (questionnaire) | one month post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Walid Habre, MD, PhD, Study Director — University of Geneva
Locations (1):
- Geneva Children's Hospital, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No